CLINICAL TRIAL: NCT00806273
Title: An in Vivo Comparison of the Debridement Efficacy of Needle Irrigation and Ultrasonic Root Canal Irrigation Techniques
Brief Title: An in Vivo Comparison of the Debridement Efficiency of Needle Irrigation Versus Ultrasonic Irrigation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Manufacturer changed device so no study will be done; ie it was never started
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00004769
Record Dates: First submitted 2008-12-08; First posted 2008-12-10 (Estimated); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Extirpation of the Tooth Pulp
Keywords: debridement; root canal

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 2 (Active Comparator): For Group II, the ultrasonic irrigation system involves using an initial irrigation with a conventional syringe followed by ultrasonic irrigation.
  Interventions: Device: Vista Ultrasonic Bleach Bypass System
- Group 1 (Active Comparator): For Group I, needle irrigation will be delivered into the pulp chamber using a syringe tip placed above the access opening and removed with high volume suction.
  Interventions: Device: Needle Irrigation

INTERVENTIONS:
Device: Vista Ultrasonic Bleach Bypass System — The ultrasonic needle will be activated by depressing the foot pedal which will begin the debridement process. Irrigants will be delivered constantly at the recommended rate via the syringe pump and the needle tip will be moved up and down with a 2mm amplitude for the entire 1 minute activation cycle, which will deliver a total of 3ml of irrigant. The ultrasonic unit will be turned off and the needle will be withdrawn from the canal.
  Arms: Group 2
Device: Needle Irrigation — irrigation with 3ml 6% NaOCl is performed moving the needle from just short of binding to 2mm coronal in constant motion for 60 seconds and left untouched in a full canal for 60 seconds.
  Arms: Group 1

SUMMARY:
Study/Protocol Title: An in vivo comparison of the debridement efficacy of needle irrigation and ultrasonic root canal irrigation techniques

1. The purpose of this study is to compare the Vista ultrasonic bypass system and conventional needle irrigation to effectively clean the bottom third of the root canal during root canal therapy.
2. Participants will be recruited from the general patient pool of the OHSU School of Dentistry. Patients will have to qualify for the study by meeting the following criteria: age between 18 and 75 years old, ASA status I or II, are currently planning treatment for the extraction of teeth, and the patient understands and signs the consent form. The principal investigator will conduct an interview with the patient and the student-provider, and obtain informed consent from the patient.
3. The teeth to be extracted will be numbed with local anesthetic. The teeth will be isolated with a rubber dam and disinfected. The pulp chamber will be accessed using normal dental equipment and the root canal will be cleaned and shaped using either the ultrasonic irrigation technique or needle irrigation. This is the first step of standard root canal therapy. The tooth will then be extracted and the principal investigator will retain extracted teeth to perform further examination to see how thoroughly the root canals were cleaned. The teeth will be discarded after study.
4. Not applicable
5. The investigational device (Vista ultrasonic bypass system) consists of a 30 gauge slot needle which attaches to an ultrasonic unit (Satalec P5). Irrigants will be delivered to the apical 1/3 of the root canal through the needle at the same time the needle is being activated ultrasonically. Irrigant delivery will be controlled by a standard syringe pump. Conventional needle irrigation will be delivered using a 27guage slot needle placed into the root canal. Irrigants will be expressed with positive pressure at a location in the canal short of the needle binding
6. Once the first step of root canal therapy has been completed, the tooth will be extracted, decalcified, and tissue specimens will be taken from the bottom 3 mm. These sections will be evaluated under magnification and remaining debris in the root canal will be quantified using the NIH Image software. The data will be statistically analyzed to determine and differences between the two irrigation techniques.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1
* ASA 2
* Pts have current treatment plan at OHSU for extraction of some or all of remaining teeth and scheduled for delivery of a removable appliance post extraction
* Teeth used are able to be isolated with rubber dam
* Understand and sign consent form

Exclusion Criteria:

* ASA 3+
* No current treatment plan at OHSU
* Severely carious teeth resulting in inability to isolate for procedure
* Unable to understand or sign consent form

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-01; Primary Completion 2009-11 (Estimated); Study Completion 2009-11 (Estimated)

PRIMARY OUTCOMES:
Software program to quantify the amount of debris left in the canals. Debris was reported as percent of canal space | 7-10 days post extraction

CONTACTS AND LOCATIONS:
Overall Officials: Craig Baumgartner, DDS, PhD, Principal Investigator — Oregon Health & Science University: Grad Endodontology